CLINICAL TRIAL: NCT04637165
Title: Exploring the Immunology of Sarcoidosis
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of York (Other)
Responsible Party: Sponsor
Other Study IDs: R2421
Record Dates: First submitted 2020-10-26; First posted 2020-11-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Sarcoidosis
Keywords: macrophage; lymphocyte; cytokine; immunology
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is a non-interventional study — This is a non-interventional study

SUMMARY:
In sarcoidosis, over activity of parts of the immune system drives the accumulation of granulomas (collections of immune cells) in affected parts of the body. To facilitate development of effective and safe treatment options in the future it will be vital to understand how and why the immune system becomes over active. The aim of this research is to work towards this goal by studying cells of the immune system and the molecular pathways inside these cells that control how they behave. This will be achieved by analysing patterns of proteins and RNA (the code used to tell cells which proteins to produce) in immune cells present in blood samples and tissue biopsies from people with sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 85 years of age, inclusive
2. Able to provide written informed consent
3. Clinician diagnosis of sarcoidosis
4. Treatment-naïve or receiving immunomodulatory therapy.

Exclusion Criteria:

1. Evidence of acute bacterial infection or other condition likely in the opinion of the investigator to significantly impact results of blood assays.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sarcoidosis
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Transcriptomics (RNA) -tissue | 3 years
  RNA expression and distribution (on different cell types) will be scored quantitatively or semi-quantitatively. Statistical analysis will be descriptive with heat maps for RNA expression (clustered using complete-linkage clustering) and charts (median and interquartile ranges) for comparisons.

SECONDARY OUTCOMES:
Protein - tissue | 3 years
  Expression and distribution (on different cell types) of proteins which will be scored quantitatively or semi-quantitatively. Results will be descriptive. Comparisons will be made using appropriate statistical techniques.
Transcriptomics (RNA) - blood | 3 years
  RNA expression in unstimulated and stimulated blood samples using Nanostring transcriptomics. Statistical analysis will be descriptive with heat maps for RNA and protein expression (clustered using complete-linkage clustering) and charts (median and interquartile ranges) for comparisons.
Cytokines - blood | 3 years
  Inflammatory mediator concentrations in unstimulated and stimulated blood samples.

OTHER OUTCOMES:
Antibodies - blood | 3 years
  Exploratory description of immunogenic proteins identified by serological analysis of recombinant complementary deoxyribonucleic acid expression libraries.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Cottingham, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No